CLINICAL TRIAL: NCT05943990
Title: Assessment of Safety and Recommended Phase 2 Dose of Autologous T Cells Engineered With an Affinity-enhanced TCR Targeting NY ESO 1 and LAGE 1a, and Co-expressing the dnTGF-βRII (GSK3845097) in Participants With NY ESO 1 and/or LAGE 1a Positive Previously Treated Advanced (Metastatic or Unresectable) Synovial Sarcoma and Myxoid/Round Cell Liposarcoma
Brief Title: Study of GSK3845097 in Previously Treated Participants With Advanced Synovial Sarcoma and Myxoid/Round Cell Liposarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in GSK's R&D priorities.
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209012 Substudy 2; 2019-004446-14 (EudraCT Number)
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: Adoptive T-cell therapy; Advanced synovial sarcoma; Advanced Myxoid/Round Cell Liposarcoma; Advanced tumors; GSK3845097; T cell receptor; Leukapheresis
MeSH Terms: conditions — Neoplasms; Liposarcoma, Myxoid | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK3845097 (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive high dose of GSK3845097 after completing lymphodepleting chemotherapy. The first study participant receiving GSK3845097 will receive the total assigned dose as 2 separate infusions 7 days apart, in aliquots of 30% (first infusion) and 70% (second infusion) of the total target dose , respectively. Based on the dose limiting toxicities reported in the first participant, then all subsequent participants treated with GSK3845097 will receive the full dose as a single, i.e., one-time, infusion.
  Interventions: Drug: GSK3845097; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: GSK3845097 — GSK3845097 was administered.
Drug: Cyclophosphamide — Cyclophosphamide was administered as lymphodepleting chemotherapy.
Drug: Fludarabine — Fludarabine was administered as lymphodepleting chemotherapy.

SUMMARY:
To assess the safety, tolerability and determine recommended phase 2 dose (RP2D) of GSK3845097 in HLA-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 positive participants with New York esophageal squamous cell carcinoma (NY-ESO)-1 and/or Cancer testis antigen 2 (LAGE-1a) positive, previously treated, advanced (metastatic or unresectable) Synovial Sarcoma (SS) and Myxoid/Round Cell Liposarcoma (MRCLS).

DETAILED DESCRIPTION:
This study is a substudy of the Master record - (209012) NCT04526509.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be >=18 years of age and weighs ≥40 kg on the day of signing informed consent
* Participant must be positive for HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 alleles
* Participant's tumor must have tested positive for NY-ESO-1 and/or LAGE-1a expression by a GSK designated laboratory
* Performance status: Eastern Cooperative Oncology Group of 0-1
* Participant must have adequate organ function and blood cell counts 7 days prior to leukapheresis
* Participant must have measurable disease according to RECIST v1.1.
* Participant has advanced (metastatic or unresectable) SS or MRCLS confirmed by local histopathology with evidence of disease-specific translocation
* Participant has completed at least one standard of care (SOC) treatment including anthracycline containing regimen unless intolerant to or ineligible to receive the therapy.
* Participants who are not candidates to receive anthracycline should have received ifosfamide unless also intolerant to or ineligible to receive ifosfamide. Participants who received neoadjuvant/adjuvant anthracycline or ifosfamide based therapy and progressed will be eligible

Exclusion Criteria:

* Central nervous system (CNS) metastases, with certain exceptions for CNS metastases in NSCLC as specified in the protocol
* Any other prior malignancy that is not in complete remission
* Clinically significant systemic illness
* Prior or active demyelinating disease
* History of chronic or recurrent (within the last year prior to leukapheresis) severe autoimmune or immune mediated disease requiring steroids or other immunosuppressive treatments
* Previous treatment with genetically engineered NY-ESO-1-specific T cells, NY-ESO-1 vaccine or NY-ESO-1 targeting antibody
* Prior gene therapy using an integrating vector
* Previous allogeneic hematopoietic stem cell transplant within the last 5 years or solid organ transplant
* Washout periods for prior radiotherapy and systemic chemotherapy must be followed
* Major surgery within 4 weeks prior to lymphodepletion
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adaptimmune Patient Enquiries, Principal Investigator — Adaptimmune
Locations (20):
- United States (11):
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Melbourne, Victoria, Australia
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: http://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a sub study of the master protocol (NCT04526509). This sub study was terminated due to a change in GSK's R&D priorities.
Groups:
- GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 1 × 10^9 - 8 × 10^9 cells of GSK3845097 as an intravenous (IV) infusion in two aliquots (approximately 30% on Day 1 and approximately 70% on Day 8) for sentinel participants or all at once on Day 1 for all other participants after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 0.1 × 10^9 - 0.8 × 10^9 cells of GSK3845097 as an intravenous (IV) infusion on Day 1 after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- No Treatment: No Treatment arm consists of participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy and T cell infusion.
Period: Overall Study
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | No Treatment
Started | 2 | 2 | 1
Completed (Participants who received T cell infusion and were followed up in this study until death or until transfer to the separate long term follow-up study are considered to have completed.) | 2 (2 participants were transferred to separate long term follow-up study 208750 (NCT03391778)) | 2 (2 participants died.) | 0
Not Completed | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | No Treatment | Total
Number analyzed (Participants) | 2 | 2 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (2.83) | 60.0 (9.90) | 41.0 | 43.8 (16.41)
Age, Customized [Count of Participants; unit: Participants]
  <=17 years | 0 | 0 | 0 | 0
  18-64 years | 2 | 1 | 1 | 4
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 2 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 0 | 1
  White | 1 | 2 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 0 | 1 | 1 | 2
  Sweden | 0 | 1 | 0 | 1
  United States | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT events were graded according to NCI-CTCAE v5.0. DLTs were defined as Grade (Gr) 4 (life-threatening and death) related to GSK3845097 2) Gr 3 (Severe or medically significant) at least possibly related to GSK3845097 and do not resolve to Gr <=1 (or Baseline) within 7 days from the onset of the event 3) Gr >=3 non-infectious pneumonitis not responding to oxygen supplementation and systemic steroid treatment 4) Any Gr 3 cytokine release syndrome (CRS) at least possibly related to GSK3845097 that does not improve to Gr <2 (moderate) toxicity within 7 days with or without dexamethasone 5) Any Gr 4 CRS at least possibly related to study product that does not improve to Gr <=2 (or Baseline) within 7 days 6) Any Gr 3 or greater neurotoxicity that does not resolve to Gr <=2 within 72 hours 7) Any Gr >=3 organ toxicity (exclusive of CRS toxicity) involving major organ systems that persists for >72 hours and occurs within 28 days of infusion.
Time Frame: Up to 28 days
Population: DLT Evaluable included participants in the mITT population (all ITT participants (All participants who started leukapheresis procedure) who received any dose of New York esophageal antigen-1 [NY ESO 1] specific T cells) who are part of the dose confirmation phase that either had a DLT or have completed the DLT assessment period of 28 days since last T cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Participants | 1 | 2

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs Based on Maximum Severity
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAE is defined as any untoward medical occurrence that, at any dose can result in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth or is medically significant or requires intervention to prevent one or the outcomes listed above. AEs and SAEs were graded according to NCI-CTCAE v5.0. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences; Grade 5- Death related to AE. AEs which start or worsen on or after T-cell infusion are classified as treatment emergent. SAEs are subset of AEs. Results for maximum severity grades has been presented.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population included all ITT participants (All participants who started leukapheresis procedure) who received any dose of NY ESO 1 specific T cells.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Participants
  AEs-Grade 4 | 2 | 0
  AEs-Grade 5 | 0 | 2
  SAEs-Grade 4 | 1 | 0
  SAEs-Grade 5 | 0 | 2

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events of Special Interest (AESI)
Description: An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. AESIs included events of Cytokine Release Syndrome (CRS), Haematopoietic cytopenias (including pancytopenia and aplastic anaemia), Graft versus Host Disease (GvHD), Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS), Guillain-Barre Syndrome (GBS), Pneumonitis and treatment-related inflammatory response at tumor site(s) and Neutropenia Grade 4 lasting more than or equal to 28 days. AEs which start or worsen on or after T-cell infusion are classified as treatment emergent.
Time Frame: Up to approximately 21 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Participants
  Participants with any AESI | 2 | 2
  Cytokine Release Syndrome (CRS) | 2 | 2
  Graft versus host disease | 1 | 1
  Haematopoietic cytopenias (including pancytopenia and aplastic anaemia) | 2 | 2
  Immune Effector-Cell Associated Neurotoxicity Syndrome | 1 | 1

4. Secondary Outcome: Overall Response Rate (ORR) Assessed by Investigator According to RECIST v1.1
Description: Overall response rate (ORR) defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via investigator assessment per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1 relative to the total number of participants in the analysis population. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response (CR) was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Confidence intervals (CI) were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Percentage of participants | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the interval of time (in months) from first documented evidence of the confirmed response (PR or CR) as assessed by local investigators to the date of disease progression per RECIST v1.1 or death due to any cause, among participants with a confirmed response of PR or CR. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Up to approximately 21 months
Population: Modified intent-to-treat (mITT) population. Only responders (CR or PR) by investigator assessment were included in this analysis. The participants analyzed in the arm (GSK3845097 0.1 × 10^9 - 0.8 × 10^9 cells) is 0, as there were no confirmed response of PR or CR.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 1 | 0
Months | 2.53 |

6. Secondary Outcome: Maximum Transgene Expansion (Cmax) of GSK3845097
Description: Cmax was defined as peak cell expansion during the interventional phase. Blood samples were collected to measure Cmax.
Time Frame: Up to 21 days
Population: Pharmacokinetic population included participants from the mITT population for whom at least one persistence sample was obtained, analysed, and was measurable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per microgram genomic DNA
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Copies per microgram genomic DNA | 54606.56 (139.944) | 105446.79 (74.752)

7. Secondary Outcome: Time to Cmax (Tmax) of GSK3845097
Description: Tmax was defined as time to peak cell expansion during the interventional phase. Blood samples were collected to measure Tmax.
Time Frame: Up to 21 days
Population: Pharmacokinetic population included participants from the mITT population for whom at least one persistence sample was obtained, analyzed, and was measurable.
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Days | 14.0 [7 to 21] | 10.5 [7 to 14]

8. Secondary Outcome: Area Under the Time Curve From Zero to Time 28 Days (AUC[0-28])
Description: Area under the cell expansion-time curve from first T-cell infusion to Day 28. Blood samples were collected to measure AUC (0-28 days).
Time Frame: Up to 28 days
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*copies per microgram genomic DNA
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells
Number analyzed (Participants) | 2 | 2
Days*copies per microgram genomic DNA | 730937.83 (151.154) | 1325540.63 (4.115)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 21 months.
Description: All cause mortality, SAEs and non-serious adverse events were reported for intent-to-treat (ITT) population that included all participants who started leukapheresis procedure.
Groups:
- No Treatment: No Treatment consists of participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy and T cell infusion.
Arm/Group | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells (N=2) | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells (N=2) | No Treatment (N=1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells (N=2) | GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells (N=2) | No Treatment (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 2 (2) | 0 (0)
Graft versus host disease in liver (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (4) | 0 (0)
White blood cell count decreased (Investigations) | 2 (5) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Interleukin level increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT05943990/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT05943990/SAP_001.pdf